CLINICAL TRIAL: NCT03346252
Title: The Effect of Botulinum Toxin A (BOTOX®) on Headache Attributed to TMD - An Open Label Trial
Brief Title: The Effect of Botulinum Toxin A on Headache Attributed to TMD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Yoly M. Gonzalez-Stucker, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000054
Record Dates: First submitted 2017-07-31; First posted 2017-11-17 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Secondary Headache Disorder
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Open Label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Botulinum Toxin type A (Experimental): Participants will be injected intramuscularly with total of 50 Units, 25 units of Botulinum A per temporalis muscle. The BTX injection will be prepared by dissolving 100 U vial in 2 ml of 0.9 % of Sodium Chloride (NaCl), yielding 25 U/ml. Each participant will receive 0.1 ml of BTX/NaCl mixture in 5 spots per temporalis muscle.
  Interventions: Drug: Botulinum Toxin type A

INTERVENTIONS:
Drug: Botulinum Toxin type A — All the participants meeting the inclusion criteria will be seen for a total of 4 visits and 3 phone interviews. Participants will complete a set of self-reporting questionnaires, assessing the disability associated with Headaches Attributed to TMD, and other pain-related TMD diagnoses, the impact of headaches on the quality of life, and psychosocial distress questionnaires.
  In addition, they will undergo 3 cycles of treatment, each 12 weeks apart.
  Other Names: Botox

SUMMARY:
This study will evaluate the effect of of botulinum toxin on the treatment of Headache Attributed to TMD.

DETAILED DESCRIPTION:
Temporomandibular Disorders (TMD) is a collective term, embracing a number of clinical problems that involve the masticatory muscles, the temporomandibular joint (TMJ) and the associated structures. The prime manifestation consists of pain of a persistent, recurring, or chronic nature . Pain-related TMD can affect the individual's daily activities, psychosocial functioning, and quality of life . The prevalence of TMD is about 10 % in the general population, making it the second most common musculoskeletal condition, after chronic lower back pain, that results in pain and disability . It has been estimated that the annual TMD management cost in the USA, excluding diagnostic imaging, in the last decade was approximately $4 billion.

The pathophysiology of pain-related TMD is poorly understood. However, multiple risk factors have been identified, such as, gender, pain during jaw function and palpation, oral parafunctions, other pain conditions, pain sensitivity and psychosocial characteristics. Because of its multifactorial nature, a multimodal conservative treatment approach is recommended, including patient education, behavioral management, physical therapy, pharmacotherapy, and occlusal splints.

Among the pain-related TMD conditions are "Headaches Attributed to TMD". This diagnosis has replaced "Headaches or facial pain attributed to Temporomandibular Joint (TMJ) disorder" described in the International Classification of Headache Disorders II (ICHD-2). It is characterized by pain in the temple area secondary to pain-related TMD that is modified by function and parafunction affected by jaw movement, function, or parafunction.

In general, headache treatment is either abortive or prophylactic. Abortive treatment manages acute headache and prophylactic treatment aims to reduce the frequency and severity of the attacks. Intramuscular injections with Botulinum Toxin (BTX) are used in the prophylactic treatment of migraine and tension type headaches. The mechanisms by which the analgesic effects of BTX are mediated are not fully understood. One mechanism is the inhibition of neurogenic inflammation by blocking neurotransmitter release from sensitized nociceptors, thus reducing peripheral sensitization. In vitro, BTX has been found to inhibit Calcitonin Gene-Related Peptide (CGRP), and BTX reduces the vascular response to algogenic substances such as capsaicin applied to human skin. Other potential analgesic mechanisms include retrograde transport of BTX by sensory neurons and inhibition of neurotransmitter release by their central terminals.

In recent years, BTX has also been used in the treatment of myogenous-TMD with mixed results. Two randomized controlled trials (RCTs) showed therapeutic benefits of BTX in the management of myogenous -TMD, while another 3 RCTs reported no significant effect of BTX in chronic myogenous -TMD pain. Varying patient samples, methodologies, and sample sizes may explain the differences. Additionally, the results have been compromised by poor methodologies, such as insufficiently powered clinical trials, and open-labeled studies. More recently, a systematic review of randomized controlled trials concluded that no consensus could be reached on the therapeutic benefit of BTX on TMD. More so, no trial on the effectiveness of BTX on the prophylactic treatment of headaches attributed to TMD has been reported to date.

The purpose of this study is to determine the effectiveness of Botulinum toxin - A in the management of headaches attributed to TMD.

Study Design The study will be carried out in the clinics of TMD and Orofacial Pain, School of Dental Medicine, University at Buffalo. A prospective open label design will be used to assess the effectiveness of BTX in the management of Headaches Attributed to TMD.

Recruitment will be done through advertising throughout the clinic and the community.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 74 years old.
* Participants with Headaches Attributed to TMD based on Diagnostic Criteria for TMD (DC-TMD) criteria.
* A minimum of 15 headaches/events per month, for the last 3 months.
* Average pain intensity in the last month of ≥5 (0 to 10 scale) where 0 is no pain and 10 is the worst pain ever.

Exclusion Criteria:

* Pregnancy
* Participants with a history of neurological/neuromuscular disorders and bleeding disorders.
* Participants taking prescribed analgesics, muscle relaxants, amino glycosides, or anticholinesterases.
* Participants currently under BTX treatment.
* Participants currently under active treatment for TMD during the last month, which includes physical therapy and pharmacological management.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Restricted to female due to: a) higher prevalence of the condition in this group and b) small sample size
Enrollment: 20 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Reduction in number of Headaches Attributed to TMD (HA) | Every 12 weeks up to 1 year
  Self-report
Reduction in Headache Impact Test-6 score (HIT-6) | Every 12 weeks up to 1 year
  Self-report.
Pressure Pain Threshold | Every 12 weeks up to 1 year
  Using algometer at the temporalis and masseter muscles

SECONDARY OUTCOMES:
Graded Chronic Pain Scale (GCPS), 1 and 6 months score | Every 12 weeks up to 1 year
  This scale provides the characterization of chronic pain as well as disability associated to the chronic pain. This scale includes 3 items for pain intensity and 4 items for function, one item for number of days of pain.
  Characteristic Pain Intensity (CPI): compute mean of items 2-4(pain right now, worst pain, average pain), and multiply by 10.
  Interference Score: compute mean of items 6-8 (daily activities, social activities, work activities), and multiply by 10.
  Interpretation Determination of Chronic Pain Grade Grade 0: (no pain, no disability)
  I Low intensity pain, without disability: (Less than 50 points in CPI and less than 3 point in disability)
  II: High Intensity pain, without disability: (Greater than or equal to 50 points in CPI and less than 3 point in disability
  III: Moderately limiting: N/A in CPI and 3-4 points in disability
  IV: Severely limiting: N/A in CPI and 5-6 points in disability
Jaw Functional Limitation Scale | Every 12 weeks up to 1 year
  Comprised within a 20-item instrument. a single global score of "jaw functional limitation" can be computed as the mean of the available items. Sub-scale scores for each type of functional limitation are computed, as follows: Mastication: mean of items 1-6. Mobility: mean of items 7-10. Verbal and non-verbal communication: mean of items 13-20. Norms have not yet been established for this instrument.
Migraine Disability Assessment/ HA-TMD | Every 12 weeks up to 1 year
  This self reported instruments comprise 6 items and based on the number of days of disability a MIDAS level is calculated as follows:
  0 to 5- MIDAS Grade I, Little or no disability 6 to 10- MIDAS Grade II, Mild disability 11 to 20- MIDAS Grade III, Moderate disability 21+ MIDAS Grade IV, Severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Yoly M Gonzalez-Stucker, DDS, MS, MPH, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784